CLINICAL TRIAL: NCT04742816
Title: Renal Effects of Hormones/Biomarkers in Transgender PrEP Recipients Sub-Study
Brief Title: Renal Effects of Hormones/Biomarkers in Transgender PrEP Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Nimish Patel, Assoc Prof Clinical, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CCTG 605s
Record Dates: First submitted 2021-01-25; First posted 2021-02-08 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Transgender; Renal Function; Hormone Replacement Therapy
MeSH Terms: interventions — Iohexol

STUDY DESIGN:
Intervention Model Description: iohexol
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Iohexol injection (Other): The research pharmacist will prepare the iohexol injection in a 1cc tuberculin syringe, consisting of 0.5cc sterile water for injection (SWFI) and 0.5cc iohexol (Omnipaque 300). The study coordinator/personnel (licensed RN) will inject the iohexol dose into the subcutaneous tissue on the opposite arm used for blood sampling; the time will be recorded. The participant will be monitored for adverse events 30 minutes post iohexol administration at the AVRC. If the participant has not had any adverse event within 30 minutes, they will be asked to leave the AVRC and return within 2 hours and 55 minutes post Iohexol injection for lab collection.
  Interventions: Diagnostic Test: IHX-CL measurements; Drug: Iohexol

INTERVENTIONS:
Diagnostic Test: IHX-CL measurements — The distribution of measured IHX-CL values and other continuous variables will be assessed to ensure a parametric distribution.
  Other Names: OMNIPAQUE; Iohexol
Drug: Iohexol — Iohexol clearance measurement
  Other Names: OMNIPAQUE

SUMMARY:
Will use a subset of the main study cohort of transgender or non-binary individuals to evaluate the relationships between self-reported exogenous hormone use, endogenous hormone values, renal biomarkers, drug levels and directly measured renal function.

DETAILED DESCRIPTION:
This cross-sectional sub-study will use a subset of the main study cohort of transgender (TG) or non-binary (NB) individuals to evaluate the relationships between self-reported exogenous hormone use, endogenous hormone values (serum estradiol, estrone, free/total testosterone), renal biomarkers, drug levels (measured by tenofovir diphosphate, TFV-DP, and emtricitabine triphosphate, FTC-TP, on dried blood spot cards and urine) and directly measured renal function (iohexol clearance).

ELIGIBILITY:
Inclusion Criteria:

* HIV-uninfected
* Identifying as transgender or nonbinary (TG/NB)
* Age ≥ 18 years (adult)
* At risk of acquiring HIV
* Calculated creatinine clearance (CRCL) ≥ 60 mL/minute
* Taking emtricitabine/tenofovir alafenamide
* Willing to receive a small dose of iohexol
* Willing to provide 30 mL blood and a urine sample

Exclusion Criteria:

* Allergy to iohexol
* Use of concurrent medications that may interfere with iohexol such as metformin, amiodarone or beta-blockers
* Anuric or unable to produce 30 mL of urine
* Other condition that, in the opinion of the investigator, would put the participant at risk, complicate interpretation of study outcome data, or would otherwise interfere with participation or achieving the study objectives

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Iohexol clearance | Day 1
  Rate of clearance (mL/min) of iohexol from the body after a small dose is administered subcutaneously. Iohexol clearance is the gold standard for measuring kidney function.

SECONDARY OUTCOMES:
Blood concentration of tenofovir | Day 1
  Tenofovir concentrations in blood and blotted on dried blood spot cards.

CONTACTS AND LOCATIONS:
Overall Officials: Nimish Patel, PharmD, Principal Investigator — UC San Diego AntiViral Research Center (AVRC)
Locations (1):
- UC San Diego AntiViral Research Center (AVRC), San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No